CLINICAL TRIAL: NCT01830608
Title: Risk Factors for Drusen Progression
Status: Withdrawn | Type: Observational
Why Stopped: Could not find a Sponsor for the study
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Ass. Prof. Priv. Doz. Dr., Medical University of Vienna
Other Study IDs: OPHT-240912
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 300 patients with AMD

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness in the Western World. The etiology and pathogenesis of this disease remain largely unknown. In Europe about two million people suffer from AMD. According to the Age-Related Eye Disease Study (AREDS) the disease can be classified into early, intermediate and late. Early age-related macular degeneration is characterized by the presence of small or medium-sized drusen and/or retinal pigmentary abnormalities. Intermediate age-related macular degeneration is characterized by large drusen or numerous medium-size drusen and/or geographic atrophy not extending to the center of the macula. Late age-related macular degeneration can be either atrophic with extension to the macula or neovascular. The late form of the disease is associated with a pronounced loss of visual acuity.

In the recent years several studies focused on risk factors for late AMD and a recent systematic review and meta-analysis reported risk factors for AMD based on 16 studies in almost 114000 subjects. Strong and consistent associations with late AMD for found for increasing age, current cigarette smoking, previous cataract surgery, and a family history of AMD. Consistent associations between late AMD and higher body mass index, history of cardiovascular disease, hypertension and higher plasma fibrinogen were also found, but the association was weak. Inconsistent associations were found for gender, ethnicity, diabetes, iris color, history of cerebrovascular disease, serum total and HDL cholesterol and triglyceride levels.

Evidence has also accumulated that other factors influence the risk for AMD. Several genetic risk factors have been identified in the last years including genes in the alternative complement pathway and the RMS2/HTRA1 region. In addition, post-hoc analysis of data from the AREDS study has indicated that reduced intake of the omega-3 free fatty acids eicosapentaenoic acid and docsahexaenoic acid are associated with the risk of late AMD thereby supporting previous population based studies. The AREDS study also revealed that reduced intake of the macular pigment lutein and zeaxanthin may be associated with late AMD, again supporting previous population-based studies. Finally, 2 small studies indicate that reduced choroidal blood flow is associated with an increased risk of developing late AMD.

Less data are available for the progression of early or intermediate AMD and the associated risk factors. This is at least partially related to the problems in quantifying progression of drusen size and volume. In the recent years, however, significant efforts have been achieved in optical coherence tomography (OCT)-based methods for quantifying drusen progression and drusen volume. Polarization-sensitive OCT is the most promising of these approaches and will be used to quantify drusen area and volume in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women aged ≥ 50 years
* AREDS categories 2 or 3 in at least one of the eyes
* No ocular surgery within last 6 months

Exclusion Criteria:

* Late form of AMD in one or two eyes (AREDS category 4)
* Moderate or severe non-proliferative diabetic retinopathy, proliferative diabetic retinopathy
* Clinically significant macular edema
* Macular or peripheral retinal dystrophies
* Ocular surgery other than uncomplicated cataract surgery
* Opacity of the ocular media by cornea or lens or diseases, which could potentially influence scan quality

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 male and female patients with age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Drusen area and volume as measured using polarization sensitive-OCT | 3 years

SECONDARY OUTCOMES:
Visual acuity and refraction | 3 years
Choroidal blood flow | 3 years
Macular pigment optical density | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria